CLINICAL TRIAL: NCT03186170
Title: Comparison of in Vitro Fertilization Rates of Oocytes and Embryo Development Using Two Techniques of Semen Processing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Campinas, Brazil (Other)
Responsible Party: Principal Investigator, Luis Bahamondes, PhD, University of Campinas, Brazil
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Unicamp/2016/LB
Record Dates: First submitted 2017-05-22; First posted 2017-06-14 (Actual); Last update posted 2017-07-25 (Actual); Status verified 2017-07

CONDITIONS: Infertility, Female
MeSH Terms: conditions — Infertility, Female

STUDY DESIGN:
Intervention Model Description: We propose to assess one method of sperm selection based on the characteristics of spermatozoa recently introduced: Sperm Selection Assay, which used a gradient of concentration of progesterone to act as chemoatractant of spermatozoa of better quality. We will assess in vitro fertilization with two techniques (SSSA versus traditional technique of swin up) as well as embryo development.
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SSA (Experimental): The investigators propose to assess one method of sperm selection based on the characteristics of spermatozoa recently introduced: Sperm Selection Assay, which used a gradient of concentration of progesterone to act as chemoatractant of spermatozoa of better quality. We will assess in vitro fertilization with two techniques (SSA versus traditional technique of swin up) as well as embryo development.
  In this arm, the sperm selection for IVF will be performed by the new proposed technique of Sperm Selection Assay which consist to expose spermatozoa a progesterone quemoatractant Sperm selection via SSA technique
  Interventions: Other: SSA sperm selection
- control (Active Comparator): The investigators propose to assess one method of sperm selection based on the characteristics of spermatozoa recently introduced: Sperm Selection Assay, which used a gradient of concentration of progesterone to act as chemoatractant of spermatozoa of better quality. We will assess in vitro fertilization with two techniques (SSSA versus traditional technique of swin up for sperm selection) as well as embryo development.
  In this arm, the sperm selection for IVF will be the traditional swin up technique with different Percoll gradient Sperm selection via traditional swin-up
  Interventions: Other: SSA sperm selection

INTERVENTIONS:
Other: SSA sperm selection — The investigators propose to assess one method of sperm selection based on the characteristics of spermatozoa recently introduced: Sperm Selection Assay, which used a gradient of concentration of progesterone to act as chemoatractant of spermatozoa of better quality. We will assess in vitro fertilization with two techniques (SSSA versus traditional technique of swin up) as well as embryo development.

SUMMARY:
The investigators propose to assess one method of sperm selection based on the characteristics of spermatozoa recently introduced: Sperm Selection Assay, which used a gradient of concentration of progesterone to act as chemoatractant of spermatozoa of better quality. We will assess in vitro fertilization with two techniques (SSSA versus traditional technique of swin up) as well as embryo development.

DETAILED DESCRIPTION:
The project is a RCT follow the orientation of CONSORT. The investigators propose to assess one method of sperm selection based on the characteristics of spermatozoa recently introduced: Sperm Selection Assay, which used a gradient of concentration of progesterone to act as chemoatractant of spermatozoa of better quality. We will assess in vitro fertilization with two techniques (SSSA versus traditional technique of swin up) as well as embryo development.

ELIGIBILITY:
Inclusion Criteria:

* infertile women who will partcipate in an IVF programme

Exclusion Criteria:

* male factor of infertility

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2017-07-15 (Actual); Study Completion 2017-07-15 (Actual)

PRIMARY OUTCOMES:
In vitro fertilization: Rate of embryo fertilizated | two weeks
  we will asses the rate of embryo fertilizated

SECONDARY OUTCOMES:
Embryo development after IVF: Rate of embryo development | two weeks
  we will asses the rate of embryo development

CONTACTS AND LOCATIONS:
Locations (1):
- University of Campinas, Campinas, São Paulo, Brazil